CLINICAL TRIAL: NCT07341880
Title: Longitudinal Monitoring of Head Impacts in Elite Junior Ice Hockey
Acronym: DRAK-CARE
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Caen (Other)
Collaborators: INSERM UMR U1075 Comète GIP Cyceron, unicaen, Caen Normandie (Unknown)
Responsible Party: Principal Investigator, Joffrey DRIGNY, Associate Professor, Consulting Physician, University Hospital, Caen
Other Study IDs: DRAK-CARE
Record Dates: First submitted 2025-11-28; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Concussion (Diagnosis); Sport-related Concussion; Hockey Player
MeSH Terms: conditions — Brain Concussion; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young Hockey Players: Elite junior ice hockey players will be monitored over one full season. Each player will wear a helmet sensor (Bearmind) to record head impacts. Heart rate variability (Polar H10) and dual-task tests will be conducted pre-, mid-, and post-season. After any concussion, both measures will be repeated at 3 days post-injury, with dual-task testing every 3 days until return to sport. Following a severe head impact, assessments will occur 3 days post-impact.
  Interventions: Device: Head impact monitoring; Other: Heart rate variability monitoring; Other: Dual-task cognitive and motor assessment

INTERVENTIONS:
Device: Head impact monitoring — Players wear a helmet-mounted sensor (Bearmind) during games and practices to record and quantify head impacts.
Other: Heart rate variability monitoring — Players wear a Polar H10 heart rate monitor to measure heart rate variability at designated times during the season. HRV is assessed pre-, mid-, and post-season, and again 3 days after a diagnosed concussion or sever head impact to evaluate autonomic nervous system responses.
Other: Dual-task cognitive and motor assessment — Players perform a dual-task test combining cognitive and motor activities while wearing a chest-mounted sensor to capture movement and performance metrics. Assessments are conducted pre-, mid-, and post-season, 3 days after a concussion or severe impact , and every 3 days until return to sport after a concussion.

SUMMARY:
This study aims to better understand how head impacts during ice hockey affect the brain and body, especially in young athletes. Even when players do not show clear signs of concussion, these repeated impacts may cause subtle changes in the brain's structure and in how the body regulates basic functions, such as heart rhythm and attention.

This study will follow elite junior ice hockey players over the course of one full season to better understand the effects of repeated head impacts. Using a small helmet sensor (Bearmind) and video analysis, researchers will record and analyze every head impact that occurs during games and practices.

Three times during the season - before, mid-season, and after - players will complete assessments of heart rate variability (using Polar H10 monitors) and a dual-task test that measures attention and coordination.

After any diagnosed concussion, players will be reassessed with both heart rate variability and dual-task testing at 3 days post-injury. Following that, dual-task testing alone will be repeated every 3 days until return to sport. Players who experience a severe head impact, as detected by the helmet sensor, will also be evaluated 3 days after the impact with both heart rate variability and dual-task testing, even if no concussion symptoms are present.

By combining these measures, the study aims to detect early physiological and cognitive changes following head impacts, improve understanding of sub-concussive effects, and support better prevention and management strategies for young athletes.

ELIGIBILITY:
Inclusion Criteria:

* Licensed athletes from the Hockey Club of Caen, playing in the U15 or U18 teams.

Exclusion Criteria:

* Inability of the participant or their legal representative to receive study information or comply with study requirements.
* Participant or legal representative cannot be reached (in person, by phone, or by email) during the sports season.
* Refusal of the participant or their legal representative to participate in the study.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population consists of licensed junior ice hockey players from the Hockey Club of Caen, competing in the U15 and U18 categories. These athletes regularly participate in competitive games and practices throughout the season and represent a cohort of developing players exposed to repeated head impacts in a real-world sports setting.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2025-09-03 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Head impact exposure | Continuously throughout one full competitive season during all games and practices (up to 9 months)
  Head impacts will be recorded using the Bearmind helmet-mounted sensor during all games and practices over the competitive season.

SECONDARY OUTCOMES:
Heart rate variability (HRV) using a 12-minute protocol | At baseline, at mid-season (14 weeks from baseline), at end of season (up to 9 months from baseline), and within 5 days following a diagnosed concussion or severe head impact.
  HRV will be measured with the Polar H10 monitor during a standardized 12-minute protocol including three phases: resting (5 min), standing (5 min), and isometric contraction (2 min). Measures will assess autonomic nervous system responses at baseline, mid-season, post-season, and post-injury.
Dual-task cognitive and motor performance | At baseline, at mid-season (14 weeks from baseline), at end of season (up to 9 months from baseline), and within 5 days following a diagnosed concussion or severe head impact.
  A dual-task test combining cognitive and motor activities will be performed while players wear a chest-mounted sensor to capture movement accuracy and reaction metrics.
Sport Concussion Assessment Tool (SCAT6) score | At baseline, and at 1 day and 4 days post-injury following a diagnosed concussion or severe head impact.
  The Sport Concussion Assessment Tool-6 (SCAT6) will be used to evaluate concussion-related symptoms, cognitive function, and balance. Assessments will be administered under standardized conditions to monitor baseline values and post-injury recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalo-Universitaire de Caen Normandie, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: Undecided